CLINICAL TRIAL: NCT02120508
Title: Phase 2 Study of rTMS Application in Aphasic Patients Evaluated With fMRI
Brief Title: Functional Neuroimage in Assessment of Post-stroke Aphasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: vghtpe user (Other Government)
Responsible Party: Sponsor-Investigator, vghtpe user, Po-Yi Tsai, MD, Taipei Veterans General Hospital, Taiwan
Organization: Taipei Veterans General Hospital, Taiwan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201207007AC
Record Dates: First submitted 2014-04-18; First posted 2014-04-22 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Stroke; Aphasia
Keywords: stroke; aphasia; rTMS; Functional MRI; Speech training
MeSH Terms: conditions — Stroke; Aphasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Hz rTMS, real (Experimental): 1 Hz rTMS over unaffected hemisphere for 15 minutes
  Interventions: Device: rTMS
- 1Hz rTMS, sham (Sham Comparator): 1Hz sham rTMS, over unaffected hemisphere for 15 minutes
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — To test the efficacy of this specific setting.
  Other Names: Magstim, Rapid2

SUMMARY:
The substantial efficacy and the possible mechanism of repetitive transcranial magnetic stimulation (rTMS) improving language recovery remained unclear. It is hypothesized that the rTMS was associated with increased synaptic connection and neural regeneration which can be evaluated via functional neuroimage and neurofiber imaging analysis. The effect of rTMS intervention was monitored by clinical testing and neuroimaging study.

DETAILED DESCRIPTION:
2-week rTMS modulation has been proved to produce substantial clinical benefit with sham-controlled study. This trial aimed to investigate the possible mechanism and make clinical correlation.

ELIGIBILITY:
Inclusion Criteria:

* Aphasic stroke in chronic stage (over 3 months)

Exclusion Criteria:

* No seizure history, no brain surgery history, no electronic device in brain or chest, no dementia

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-08 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Concise Chinese Aphasia Test | Before the rTMS intervention, at 2nd week, and 3rd month
  Assess the linguistic skills such as conversation, expression, description, comprehension...

SECONDARY OUTCOMES:
Functional MRI | Before rTMS intervention, and at the day completing the rTMS treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Po-Yi Tsai, MD, Principal Investigator — Department of physical medicine and rehabilitation, Taipei Veterans General Hospital
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Tsai PY, Wang CP, Ko JS, Chung YM, Chang YW, Wang JX. The persistent and broadly modulating effect of inhibitory rTMS in nonfluent aphasic patients: a sham-controlled, double-blind study. Neurorehabil Neural Repair. 2014 Oct;28(8):779-87. doi: 10.1177/1545968314522710. Epub 2014 Feb 13. PMID 24526709
- [Derived] Wang CP, Hsieh CY, Tsai PY, Wang CT, Lin FG, Chan RC. Efficacy of synchronous verbal training during repetitive transcranial magnetic stimulation in patients with chronic aphasia. Stroke. 2014 Dec;45(12):3656-62. doi: 10.1161/STROKEAHA.114.007058. Epub 2014 Nov 6. PMID 25378426